CLINICAL TRIAL: NCT06506617
Title: HCAPPED I: HCAP - Pcr in Emergency Department. Early Multiplex PCR on Respiratory Samples From Patients With Pneumonia. A No-profit Observation Prospective Study
Brief Title: HCAPPED I: HCAP-Pcr in Emergency Department
Acronym: HCAPPED-I
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: CEAVC 26198_oss
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Pneumonia; Bronchoalveolar Lavage; Antimicrobial Treatment; Sputum
Keywords: Bronchoalveolar lavage; Endotracheal Aspirate; Antimicrobial treatment; pneumonia; hcap; pcr multiplex; moleculas syndromic panel; bal; bas; eta; sputum
MeSH Terms: conditions — Pneumonia; De Lange Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — BAL, BAS, ETA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCR multiplex (BIOFIRE® FILMARRAY® Pneumonia plus Panel): The study seeks to assess the utility of molecular diagnostic tests in the emergency department for the microbiological etiological diagnosis of healthcare-associated pneumonia (HCAP).
  In clinical practice, patients with respiratory and infectious symptoms undergo blood sample collection for blood gas, chemical-physical, and culture analyses, urine samples for urinary antigen testing, and imaging diagnostics (X-ray, CT, ultrasound). Due to local infection control and surveillance measures, all patients with respiratory symptoms undergo a nasopharyngeal antigen test for SARS-CoV-2 as part of standard clinical practice.
  After completing the diagnostic work-up and diagnosing HCAP pneumonia, endobronchial samples are typically collected for multiplex PCR testing (BIOFIRE® FILMARRAY® Pneumonia plus Panel). Patients from whom these samples are collected are those needing high-flow oxygen therapy (VM35 or FiO2 higher, Reservoir, HFNC, NIV, CPAP), undergoing IOT, SOFA ≥2, PaO2/FiO2 < 200, o

SUMMARY:
Prospective Observational Study (on Diagnostic Procedure) - Single-Center, Non-Profit.

A pilot study will be conducted on a prospective cohort of patients with HCAP (Healthcare-Associated Pneumonia). This study will be conducted on a single arm of patients. No control group or randomization is planned.

The use of syndromic molecular panels in pneumonias with risk factors for MDR (multidrug-resistant) pathogens, such as in patients with HCAP, has become common practice. However, the use of this tool is reserved for patients with severe forms of HCAP (PIRO>2, at least moderate ARDS, and respiratory failure requiring high-flow oxygen during sepsis) (30), and it is not yet standardized by international guidelines. The decision to use this tool or not is currently at the clinician's discretion and is usually reserved for the severe forms mentioned above. The study aims to determine if the early use of this tool has a real benefit on the management of antibiotic therapy for these patients in terms of therapeutic changes compared to corporate and international guidelines.

Duration of patient enrollment: 1 year. Duration of the study: 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

All patients over the age of 18 who undergo bronchoalveolar lavage (BAL) in the Emergency Department (DEA), with a Rankin score of less than 5, and who are admitted to the Emergency Department with a diagnosis of healthcare-associated pneumonia (HCAP) of bacterial, viral, or fungal origin. The diagnosis must be confirmed by clinical and radiological criteria according to the IDSA guidelines, which include: New pulmonary infiltrate on chest X-ray, Evidence that the infiltrate is of infectious origin, At least two of the following three clinical signs: Fever higher than 38 °C, Leukocytosis or leukopenia, Purulent secretions.

Additionally, patients must meet at least one of the following criteria:

* Need for high-flow oxygen therapy (VM35 or FiO2 >35%, Reservoir, HFNC, NIV, CPAP)
* Intubation (IOT)
* SOFA score ≥2 or PSI score >85 (age 75 + IR)
* Horowitz index (PaO2/FiO2) < 200

Exclusion Criteria:

* Lack of consent
* Age under 18 or over 90
* Pregnancy
* Life expectancy less than 3 months
* Hospital admission >48 hours (hospital-acquired pneumonia - HAP)
* Rankin score ≥ 5
* Community-acquired pneumonia (CAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 who undergo bronchoalveolar lavage (BAL) in the Emergency Department (DEA), with a Rankin score of less than 5, and who are admitted to the Emergency Department with a diagnosis of healthcare-associated pneumonia (HCAP) of bacterial, viral, or fungal origin.
  A patient is considered to have HCAP if they meet any of the following conditions:
  Hospitalized in an acute care hospital for two or more days within 90 days of symptom onset Residing in a nursing home or long-term care facility Received intravenous antibiotic therapy, chemotherapy, or wound care within the past 30 days Attended a hospital or hemodialysis clinic within the past 30 days for medical reasons, visits, or day services
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-07-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
evaluate the impact of early use of multiplex PCR | perioperatively/periprocedurally
  The primary objective of the study is to evaluate the impact of early use of multiplex PCR on empirical antibiotic therapy. This will be measured by considering the percentage of cases in which the use of multiplex PCR alters the therapy ('escalation' and 'de-escalation') compared to local empirical antibiotic therapy guidelines within 24 hours of hospital admission.

SECONDARY OUTCOMES:
Time to Antibiotic Escalation or De-escalation | up to 3 months
  Measure the time from hospital admission to the escalation or de-escalation of antibiotic therapy.
Length of Hospital Stay | up to 3 months
  Assess the total duration of the hospital stay.
Need for Escalation of Supportive Therapy: | up to 3 months
  Evaluate the necessity for increased supportive therapy, defined as: a) Need for invasive or non-invasive ventilation b) Transfer to a higher level of care c) In-hospital mortality from any cause (complicated course)
Duration of Antibiotic Therapy: | up to 3 months
  Track the length of time antibiotics are administered.
De-escalation of Antibiotic Therapy | 7 days from admission
  Assess the de-escalation of antibiotic therapy within the first 7 days of inclusion in the study.
Escalation of Antibiotic Therapy | 7 days from admission
  Assess the escalation of antibiotic therapy within the first 7 days of inclusion in the study.
Identification of HCAP Etiology | 7 days from admission
  Determine the cause of HCAP within the first 7 days of inclusion using all methods: multiplex PCR, culture tests, antigen detection, and serology.
In-hospital Mortality | up to 3 months
  Measure in-hospital mortality rates for pneumonia and all causes.
30-day Mortality and Readmission | 30 days from discharge
  Measure mortality rates for pneumonia and all causes, and track readmissions within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Pelagatti Lorenzo, Dr, Principal Investigator — AOU Careggi
Locations (1):
- Azienda ospedaliero universitaria careggi, Florence, Tuscany/Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided